CLINICAL TRIAL: NCT02857712
Title: Phase II Study on Inlyta® (Axitinib) in Recurrent and/or Metastatic Salivary Gland Cancers (SGCs) of the Upper Aerodigestive Tract
Brief Title: Axitinib in R/M Salivary Gland Cancers of the Upper Aerodigestive Tract - SGC-AX14
Acronym: SGC-AX14
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INT 135/14
Record Dates: First submitted 2016-05-06; First posted 2016-08-05 (Estimated); Last update posted 2019-08-30 (Actual); Status verified 2019-08

CONDITIONS: Salivary Gland Cancers
MeSH Terms: conditions — Salivary Gland Neoplasms | interventions — Axitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Axitinib (Experimental): Axitinib will be administered at 5 mg BID (starting dose); in case of no adverse events above CTCAE version 4.0 Grade 2 for a consecutive 2-week periods, the dose may be increased to 7 mg BID and further to 10 mg BID using the same criteria until tumor progression, unacceptable toxicity or other criteria for discontinuation is met.
  Interventions: Drug: Axitinib

INTERVENTIONS:
Drug: Axitinib — Axitinib will be self orally administered at 5 mg twice daily approximately every 12 hours, on a continuous basis (each morning and evening), in 4 week cycles until tumour progression, unacceptable toxicity or other criteria for discontinuation is met. Patients who tolerate axitinib with no adverse events axitinib-related should have a dose increased until to 10 mg twice.
  Other Names: Inlyta

SUMMARY:
SGCs are rare (less than 1% of head and neck cancers) and include many malignant histotypes. SGCs are treated mainly with surgery, followed by radiotherapy in selected cases. Chemotherapy is reserved for palliative treatment of metastases or local recurrence but results in term of response rate are very low. Adenoid cystic cancer (ACC) is the most common SGC histotype observed in metastatic subjects while the other histotypes (non-ACC) such as mucoepidermoid cancer (MEC), salivary duct gland cancer, adenocarcinoma, myoepithelial carcinoma are more uncommon. A phase II trial with sorafenib carried out in 37 subjects (19 ACC and 18 non-ACC) with recurrent and/or metastatic SGCs showed a response rate of 16% (11% in ACC and 22% in non-ACC). In preclinical models, VEGF seems to contribute to tumor aggressiveness and to distant metastatization of SGCs, in particular in ACC and MEC. Remarkably three confirmed partial responses, one ACC, one renal cancer and one lung cancer, on 36 patients were observed in a phase I study with Inlyta, a potent VEGFR specific-inhibitor approved by FDA as second line treatment for renal cancer. Based on these data, we want to test Inlyta in patients with relapsed and/or metastatic SGC.

DETAILED DESCRIPTION:
Carcinomas of the salivary glands (SGCs) are rare, (less than 1% of all cancers of the head and neck and include more than 20 malignant histotypes). They can occur both in major and minor salivary glands, are locally aggressive, demonstrating invasiveness that leads to involvement of the facial nerve, skin, bone and surrounding soft tissue. The standard treatment is surgical excision, followed by radiotherapy in selected cases such as high-grade histotypes, advanced disease and neck nodes diffusion. Loco-regional recurrence occurs in 16% to 85%, it can be managed in very selected cases with further surgery and/or radiotherapy, although the prognosis of these patients remains poor. Adenoid cystic cancer (ACC) is the most common SGC histotype observed in metastatic subjects (60%), while the other histotypes (non-ACC) such as mucoepidermoid cancer (MEC), salivary duct gland cancer, adenocarcinoma, myoepithelial carcinoma are more uncommon. Distant metastases are the principal cause of failure, being diagnosed in 25-55% of the patients. Only 20% of the patients with distant metastases is alive at 5 years. First-line treatment is palliative chemotherapy that is typically not associated with solid data showing any benefit neither in response rate nor in outcome. Very recently a phase II trial with sorafenib has been carried out in 37 subjects (19 ACC and 18 non-ACC) with recurrent and/or metastatic SGCs. Interestingly, a response rate of 16% (95% CI 6,2-32,0) was observed, 11% in ACC and 22% in non-ACC cases with two outstanding responses in patients with an high-grade MEC. In one case the metastatic lesion evolved in a cavitation as observed with antiangiogenic agents. In preclinical models, VEGF seems to contribute to tumor aggressiveness as well as to distant metastatization of SGCs, in particular in ACC and MEC. Remarkably three confirmed partial responses, one ACC, one renal cancer and one lung cancer, on 36 patients were observed in a phase I study with Inlyta®. These results prompted a phase II study to test the activity of axitinib in relapsed and/or metastatic and progressive ACC patients. Results were 9% of partial responses and 75% of stable disease as best overall response. Inlyta®, a potent VEGFR specific-inhibitor, has been approved by FDA as second line treatment for renal cancer. Based on preclinical and clinical data, we believe that targeting VEGFR might represent a rational basis to further test Inlyta® in patients with relapsed and/or metastatic ACC but also in subjects with recurrent/metastatic non-ACC .

Open-label, monocentric, single arm phase II study evaluating the activity and safety of axitinib in recurrent and/or metastatic tumors of salivary gland. 26 patients with histologically proven relapsed or metastatic SGC, progressed within 6 months at study entry will be enrolled over two years. A 2-stage Simon design will be applied: 15 patients enrolled into step one and if a least 1/15 response is observed, 11 additional patients will be enrolled into second step. Axitinib will be administered orally at 5 mg twice daily to patients for the first two weeks. Patients who tolerate axitinib with no adverse events axitinib-related should have a dose increased until to 10 mg twice. The drug will be taken until progression of disease or intolerable toxicity. Tissue paraffin block from primary lesion or metastasis will be collected for CRTC1-MAML2 translocation analysis in MEC; MYB-NFIB translocation analysis in ACC; androgen receptor and HER2 analysis in SDC and adenocarcinoma NOS.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven relapsed and/or metastatic salivary gland cancer for which potentially curative options such as surgery or radiotherapy are not indicated.
* Archival tissue samples or unstained 20 slides from primary tumor or metastasis for translational biological research.
* Subjects with at least one uni-dimensional measurable lesion by CT-scan or MRI according to RECIST criteria 1.1 (target lesion). A previously treated lesion by radiotherapy can be chosen as target lesion only if progression in the respective lesion has been demonstrated during or following radiotherapy.
* Clinical or radiological progression of disease within 6 months at study entry. Progression of disease by RECIST is not required.
* Age ≥18 years
* ECOG Performance Status < 2
* Life expectancy of > 3 months
* Adequate bone marrow, liver and renal function as assessed by the following laboratory requirements to be conducted within 7 days prior to screening:
* Hemoglobin >9.0 g/dl
* Neutrophil count (ANC) >1,000/mm3
* Platelet count ≥ 75,000/µl
* Total bilirubin < 1.5 times the upper limit of normal
* ALT and AST < 2.5 x upper limit of normal (<5 x upper limit of normal for patients with liver metastases)
* Serum creatinine <1.5 x upper limit of normal
* Urinary protein < 2+ by urine dipstick
* Alkaline phosphatase < 4 x ULN
* PT-INR/PTT <1.5 x upper limit of normal (Patients who are being therapeutically anticoagulated with an agent such as coumadin or heparin will be allowed to participate provided that no prior evidence of underlying abnormality in these parameters exists)
* No evidence of preexisting uncontrolled hypertension as documented by 2 baseline blood pressure readings taken at least 1 hour apart. The baseline systolic blood pressure reading must be ≤140, and the baseline diastolic blood pressure readings must be < 90. Patients whose hypertension is controlled by antihypertensive therapies are eligible.
* Signed written informed consent

Exclusion Criteria:

* Symptomatic metastatic brain or meningeal tumors unless the patient is > 6 months from definitive therapy, has a negative imaging study within 4 weeks of study entry and is clinically stable with respect to the tumor at the time of study entry
* Previous systemic therapy for metastatic disease is not allowed (chemotherapy or TKI)
* History of cardiac disease: congestive heart failure >NYHA class 2; active CAD (MI more than 6 mo prior to study entry is allowed); cardiac arrhythmias requiring anti-arrhythmic therapy (beta blockers or digoxin are permitted) or uncontrolled hypertension
* Known allergic reaction to any of the components of the treatment
* Substance abuse, medical, psychological or social conditions that may interfere with the patient's participation in the study or evaluation of the study results
* Legal incapacity or limited legal capacity
* Active clinically serious infections (> grade 2 NCI-CTC version 4.0)
* Medical or psychological condition which, in the opinion of the investigator, would not enable the patient to complete the study or knowingly sign the Informed Consent
* Pregnant or breast-feeding patients. Women of childbearing potential must have a negative pregnancy test performed within 7 days of the start of treatment. Both men and women enrolled in this trial must use adequate barrier birth control measures during the course of the trial and two weeks after the completion of trial
* Previous or concurrent cancer that is distinct in primary site or histology from the cancer being evaluated in this study except cervical carcinoma in situ, treated basal cell carcinoma, superficial bladder tumors [Ta, Tis and T1] or any cancer curatively treated > 3 years prior to study entry.
* Patients with seizure disorder requiring medication (such as steroids or anti-epileptics)
* History of organ allograft.
* Patients with evidence or history of bleeding diathesis
* Gastrointestinal abnormalities (i.e. inability to take oral medication; malabsorption syndrome)
* Requirement for anticoagulant therapy with oral vitamin K antagonists
* Anticancer chemotherapy or immunotherapy during the study or within 4 weeks of study entry.
* Radiotherapy during study or within 3 weeks of start of study drug. (Palliative radiotherapy will be allowed)
* Major surgery within 2 weeks of start of study
* Use of biologic response modifiers, such as G-CSF, within 3 week of study entry [G-CSF and other hematopoietic growth factors may be used in the management of acute toxicity such as febrile neutropenia when clinically indicated or at the discretion of the investigator, however they may not be substituted for a required dose reduction; patients taking chronic erythropoietin are permitted provided no dose adjustment is undertaken within 2 months prior to the study or during the study]
* Investigational drug therapy outside of this trial during or within 4 weeks of study entry
* Current use or anticipated need for treatment with drugs inhibiting CYP3A4
* Current use or anticipated need for treatment with drugs inducing CYP3A4 or CYP1A2

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2014-12; Primary Completion 2018-10 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Objective response rate (CR+PR) | 2 years and 7 months
  Objective response rate (CR+PR) will be evaluated according to RECIST response evaluation criteria 1.1 at any subsequent re-evaluation

SECONDARY OUTCOMES:
Progression free survival | 2 years and 7 months
  PFS according to RECIST criteria 1.1
Overall survival | 2 years and 7 months
  After study drug treatment ends, patients will be contacted each 6 months to determine survival status.
Evaluation acute toxicity (according to CTCAE v4.0) | 2 years and 7 months
  Acute toxicity according to CTCAE v4.0
Duration of response | 2 years and 7 months
  The duration of response will be evaluated to assess the duration of activity of axitinib (CR+PR+SD)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Licitra, Principal Investigator — Fondazione IRCCS Istituto Nazionale dei Tumori, Milano
Locations (1):
- Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, Italy

IPD SHARING:
Plan to Share IPD: No
Only study results will be shared through publication on scientific indexed journals